CLINICAL TRIAL: NCT02559349
Title: Gut Microbiota And Radiotherapy
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15415
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Lung Tumor
Keywords: Stereotactic Body Radiotherapy; SBRT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool Sample
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Stool Collection

SUMMARY:
A pilot, single arm, single center study to determine the feasibility of obtaining stool samples from adult patients receiving SBRT to a lung tumor, if SBRT induces changes in the gut microbiota and to obtain preliminary data about possible correlation of baseline composition and changes in gut microbiota with tumor response, local control, and development of pneumonitis/other side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is planned to receive Stereotactic Body Radiotherapy (SBRT) to a lung lesion (either presumed or biopsy-proven NSCLC
* Age 18 years old or older
* Patient capable of giving informed consent

Exclusion Criteria

* Use of antibiotics, antifungal, antivirals or antiparasitics during the 4 weeks prior to registration
* Active infection with oral temperature >100°F
* Use of corticosteroids, methotrexate or immunosuppressive drugs during the 4 weeks prior to registration
* Use of chemotherapy during the 4 weeks prior to radiotherapy or during radiotherapy. Chemotherapy cannot begin before the collection of the 30-day post treatment sample (S4).
* Confirmed or suspected HIV, HBV or HCV
* Chronic constipation (bowel movements less frequent than every other day)
* Active uncontrolled gastrointestinal disorders such as inflammatory bowel disease, moderate/severe irritable bowel syndrome, persistent, infectious gastroenteritis, colitis or gastritis, persistent or chronic diarrhea of unknown etiology, Clostridium Difficile infection (recurrent) or Helicobacter Pylori infection (untreated)
* Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years. Any major bowel resection at any time
* Patients on anti-diarrheal medications
* Patients on probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving SBRT to a lung tumor
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of subject providing stool samples | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States